CLINICAL TRIAL: NCT02184429
Title: A Phase 1, Double Blind, Sponsor Open, Placebo Controlled Combined Single And Multiple Ascending Dose Study To Investigate The Safety, Tolerability And Food Effect On Pharmacokinetics Of PF-06669571 Following Oral Doses In Healthy Subjects
Brief Title: A Study To Understand Safety And Plasma Concentrations Of PF-06669571 During And Following The Oral Administration Of Single And Multiple Doses Of PF-06669571 In Healthy Volunteers Under Fasted And Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7821001
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2016-03

CONDITIONS: Healthy
Keywords: First in human; single ascending dose study; multiple ascending dose study; safety and tolerability; pharmacokinetics; food effect; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — PF-06669571

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Single Ascending Dose-1 (Experimental): Single ascending doses of PF-06669571 administered to healthy volunteers in a cross over study design
  Interventions: Drug: PF-06669571
- Single Ascending Dose-2 (Experimental): Single ascending doses of PF-06669571 administered to healthy volunteers in a cross over study design
  Interventions: Drug: PF-06669571
- Multiple Ascending Dose-1 (Experimental): Daily dose of PF-06669571 in healthy volunteers
  Interventions: Drug: PF-06669571
- Multiple Ascending Dose-2 (Experimental): Daily dose of PF-06669571 in healthy volunteers
  Interventions: Drug: PF-06669571
- Multiple Ascending Dose-3 (Experimental): Daily dose of PF-06669571 in healthy volunteers
  Interventions: Drug: PF-06669571
- Multiple Ascending Dose-4 (Experimental): Daily dose of PF-06669571 in healthy volunteers
  Interventions: Drug: PF-06669571
- Multiple Ascending Dose-5 (Experimental): Daily dose of PF-06669571 in healthy volunteers
  Interventions: Drug: PF-06669571

INTERVENTIONS:
Drug: PF-06669571 — Single ascending doses of PF-06669571 as extemporaneously prepared solution/suspension, once week in a cross over study: 0.2 mg 0.4 mg, 0.75 mg, 1.50 mg and placebo
  Arms: Single Ascending Dose-1
Drug: PF-06669571 — Single ascending doses of PF-06669571 as extemporaneously prepared solution/suspension, once week in a cross over study: 3 mg 6 mg, 10 mg, 3 mg (fed) and placebo
  Arms: Single Ascending Dose-2
Drug: PF-06669571 — Oral dosing of 0.15 mg PF-06669571 as extemporaneously prepared solution/suspension or powder in capsule formulation for 14 days
  Arms: Multiple Ascending Dose-1
Drug: PF-06669571 — Oral dosing of 0.5 mg PF-06669571 as extemporaneously prepared solution/suspension or powder in capsule formulation for 14 days
  Arms: Multiple Ascending Dose-2
Drug: PF-06669571 — Oral dosing of 1.5 mg PF-06669571 as extemporaneously prepared solution/suspension or powder in capsule formulation for 14 days. This dose may be reached by a titration scheme
  Arms: Multiple Ascending Dose-3
Drug: PF-06669571 — Oral dosing of 4.5 mg PF-06669571 as extemporaneously prepared solution/suspension or powder in capsule formulation for 14 days. This dose may be reached by a titration scheme
  Arms: Multiple Ascending Dose-4
Drug: PF-06669571 — Oral dosing of 9.0 mg PF-06669571 as extemporaneously prepared solution/suspension or powder in capsule for 14 days. This dose may be reached by a titration scheme
  Arms: Multiple Ascending Dose-5

SUMMARY:
This study is designed to evaluate the safety and plasma concentrations of PF-06669571 in healthy volunteers following single and multiple ascending doses of PF-06669571. Effect of food on PF-06669571 plasma concentrations will be be evaluated after a single dose of PF-06669571. During multiple dose phase, PF-06669571 will be administered daily for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).

Female subjects of non-childbearing potential must meet at least one of the following criteria:

1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state;
2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.

   * Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
   * Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
   * Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
* Screening supine blood pressure >= 140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of rest. If BP is >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), repeat per local standard operating procedures (SOP). If orthostatic changes are present and deemed to be clinically significant by the investigator, Subject can be excluded.
* For subjects who answer "Yes" to the Columbia Suicide Severity Rating Scale (C-SSRS) questions 4 or 5, a risk assessment should be done by a qualified mental health professional (MHP: a psychiatrist or licensed PhD level clinical psychologist) to assess whether it is safe for the subject to participate in the study. In addition, subjects deemed by the investigator to be at significant risk of suicidal or violent behavior should be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with categorical scores on the Columbia Suicide Severity Rating Scale (C-SSRS) | screening,Day 28
  C-SSRS assessed whether participant experienced following: completed suicide (1), suicide attempt (2) (response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (3)("Yes" on "preparatory acts or behavior"), suicidal ideation (4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior (7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior").

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) after single dose | 0-Day 5
  Cmax after a single dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) after single dose | 0-Day 5
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) after single dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] after single dose | 0-Day 5
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf) after single dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) after single dose | 0-Day 5
  Tmax after single dose
Plasma Decay Half-Life (t1/2) after single dose | 0-Day 5
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half after single dose
Apparent Oral Clearance (CL/F) after single dose | 0-Day 5
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood after single dose
Apparent Volume of Distribution (Vz/F) after single dose | 0-Day 5
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Maximum Observed Plasma Concentration (Cmax) on Days 1, 7 and 14 after multiple daily dose | 0-Day 18
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) on days 1,7,14 after multiple daily doses | 0-Day 18
Time to Reach Maximum Observed Plasma Concentration (Tmax) on days 1,7 14 after multiple daily doses | 0-Day 18
Apparent Oral Clearance (CL/F) on day 7 and 14 after multiple daily doses | 0-Day 18
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Pre dose concentrations (Ctrough) on days 7 and 14 after multiple daily doses | 0-Day 18
Minimum Observed Plasma Trough Concentration (Cmin) on days 7 and 14 after multiple daily doses | 0-Day 18
Accumulation ratio (Rac) for AUCtau on days 7 and 14 after multiple daily doses | 0-day 18
Accumulation ratio (Rac) for Cmax on days 7 and 14 after multiple daily doses | 0-Day 18
Plasma Decay Half-Life (t1/2) on day 14 after multiple daily doses | 0-Day 18
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Volume of Distribution (Vz/F) on day 14 after multiple daily doses | 0-Day 18
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Renal clearance (CLr) on day 14 | 0-Day 18
Amount of unchanged drug recovered in urine during the dosing interval (AEtau) on Day 14 after multiple daily doses | 0-Day 18
Percent of dose recovered unchanged in urine during the dosing interval (AEtau%) on Day 14 after multiple daily doses | 0-Day 18
Peak to Trough ratio at Steady State (PTR) | 0-Day 18
  Cmax to Cmin ratio at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7821001&StudyName=A%20Study%20To%20Understand%20Safety%20And%20Plasma%20Concentrations%20Of%20PF-06669571%20During%20And%20Following%20The%20Oral%20Administration%20Of%20Single%20And%20Multipl